CLINICAL TRIAL: NCT05087056
Title: A Phase IIb, Randomized, Observer-Blind Study to Describe the Safety, Tolerability, and Immunogenicity of MenABCWY Administered on Different Dosing Schedules in Healthy Adolescents
Brief Title: Safety, Tolerability, and Immunogenicity of MenABCWY Administered on Different Dosing Schedules in Healthy Adolescents
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 215344; 2021-001670-33 (EudraCT Number)
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Meningitis, Meningococcal
Keywords: MenABCWY; Safety; Tolerability; Immunogenicity; Healthy adolescents; Invasive meningococcal disease
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind study. Participants and study evaluators will be unaware of vaccine administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABCWY-24 Group (Experimental): Participants receive 2 doses of the MenABCWY vaccine at Day 1 and Day 721, 1 dose of Placebo at Day 1441.
  Interventions: Combination Product: MenABCWY vaccine; Combination Product: Placebo
- ABCWY-48 Group (Experimental): Participants receive 2 doses of the MenABCWY vaccine at Day 1 and Day 1441, 1 dose of Placebo at Day 721.
  Interventions: Combination Product: MenABCWY vaccine; Combination Product: Placebo

INTERVENTIONS:
Combination Product: MenABCWY vaccine — Two doses of the MenABCWY vaccine, administered intramuscularly in the deltoid region of the non-dominant arm, on a 0-, 24-month schedule in the ABCWY-24 Group, and a 0-, 48-month schedule in the ABCWY-48 Group.
Combination Product: Placebo — Single dose of Placebo (saline solution in pre-filled syringe), administered intramuscularly in the deltoid region of the non-dominant arm, at Day 1441 in the ABCWY-24 Group, and at Day 721 in the ABCWY-48 Group.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and immunogenicity of the combined meningococcal groups A, B, C, W and Y (MenABCWY) vaccine (GSK3536819A) intended to protect against invasive meningococcal disease (IMD) caused by all 5 meningococcal serogroups.

ELIGIBILITY:
Inclusion Criteria:

* Participants or/and participants' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant/parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* Written informed assent obtained from the participant (if applicable) prior to performing any study specific procedure.
* A male or female between, and including, 11 and 14 years of age (i.e. 14 years + 364 days) at the time of the first vaccination.
* Healthy participants as established by medical history, physical examination and clinical judgment of the investigator before entering into the study.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, hysterectomy, bilateral-salpingectomy or bilateral ovariectomy.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 30 days prior to first vaccination, and
  * has a negative pregnancy test* on the day of vaccination, and
  * has agreed to follow adequate contraception for 30 days before each of the 2 subsequent vaccinations and for 30 days after each vaccination * Urine samples for pregnancy testing will be collected from female participants of childbearing potential at Visit 1, Visit 3 and Visit 5 prior to the vaccination.

Exclusion Criteria:

Medical conditions

* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection within 60 days of enrolment.
* Progressive, unstable or uncontrolled clinical conditions.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any neuroinflammatory, congenital neurological conditions, encephalopathies, seizures. History of febrile convulsions should not lead to exclusion.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s)/product(s).

  * Hypersensitivity, including allergy, to any component of vaccines, including diphtheria toxoid (CRM197) and latex medicinal products or medical equipment whose use is foreseen in this study.
* Abnormal function or modification of the immune system resulting from:

  * Autoimmune disorders or immunodeficiency syndromes.
  * Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 90 days prior to study vaccination. This will mean prednisone equivalent ≥20 mg/day for adult participants / ≥0.5 mg/kg/day with maximum 20 mg/day for paediatric participants. Inhaled and topical steroids are allowed.
  * Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to study vaccination.
  * Administration of long-acting immune-modifying drugs at any time during the study period.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study vaccine(s)/product(s) during the period starting 30 days before the first dose of study vaccine(s)/product(s) (Day -29 to Day 1), or planned use during the study period.
* Previous vaccination with any meningococcal (MenB or MenACWY) vaccine at any time prior to informed consent/ assent (as applicable) with the exception of meningococcal C (conjugated or polysaccharide) vaccination, if the last dose of MenC was received at ≤24 months of age.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the administration of study vaccine/product or planned administration before the next blood sampling visit.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first vaccine/product dose(s). For corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants / ≥0.5 mg/kg/day with maximum of 20 mg/day for paediatric participants. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or medical device).

Other exclusions

* Child in care.
* Pregnant or lactating female.
* Female planning to become pregnant / planning to discontinue contraceptive precautions during the windows reported in the inclusion criterion.
* History of /current chronic alcohol abuse and/or drug abuse as determined by the investigator.
* Any study personnel or immediate dependants, family, or household members.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with human serum bactericidal assay (hSBA) titers ≥ lower limit of quantitation (LLOQ) for each N. meningitidis serogroup B indicator strains | At Baseline (Day 1)
  The immune response to 2 doses of the MenABCWY vaccine administered on a 0-, 24-month schedule, and a 0-, 48-month schedule is evaluated against each N. meningitidis serogroup B indicator strains.
Percentage of participants with hSBA titers ≥ LLOQ for each N. meningitidis serogroup B indicator strains | At 1 month after the second dose of MenABCWY (Day 751 for the ABCWY-24 Group and Day 1471 for the ABCWY-48 Group)
  The immune response to 2 doses of the MenABCWY vaccine administered on a 0-, 24-month schedule, and a 0-, 48-month schedule is evaluated against each N. meningitidis serogroup B indicator strains.
Percentage of participants with solicited administration site events | During the 7 days (including the day of vaccination) following each vaccination (Vaccines administered at Day 1, Day 721 and Day 1441)
  The solicited administration site events include pain, redness, swelling and induration. Redness, swelling, and induration are summarized according to defined severity grading scales: None (0 to 24mm); Mild (25 to 50mm); Moderate (51 to 100mm); Severe (>100mm). Injection site pain is summarized according to "mild", "moderate" or "severe".
Percentage of participants with solicited systemic events | During the 7 days (including the day of vaccination) following each vaccination (Vaccines administered at Day 1, Day 721 and Day 1441)
  The solicited systemic events include fever, headache, nausea, myalgia, arthralgia and fatigue. Fever is defined as body temperature 38.0°C (100.4°F). The preferred location for measuring temperature in this study is the oral route. Solicited systemic events (except fever) are summarized according to "mild", "moderate" or "severe".
Percentage of participants with any unsolicited adverse events (AEs) including all serious adverse events (SAEs), AEs leading to withdrawal, adverse events of special interest (AESIs) and medically attended AEs | During the 30 days (including the day of vaccination) following each vaccination (Vaccines administered at Day 1, Day 721 and Day 1441)
  An unsolicited AE is an AE that was not included in a list of solicited events and must have been spontaneously communicated by a participant/participant's parent(s)/ Legally Acceptable Representative(s) who has signed the informed consent. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject or is an abnormal pregnancy outcome. AESIs are predefined AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterise and understand it. Medically attended AEs are symptoms or illnesses requiring a hospitalisation, or an emergency room visit, or visit to/by a health care provider.
Percentage of participants with SAEs, AEs leading to withdrawal, AESIs and medically attended AEs | During the 6 months (including the day of vaccination) following the first vaccination (Vaccine administered at Day 1)
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject or is an abnormal pregnancy outcome. AESIs are predefined (serious or non-serious) AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterise and understand it. Medically attended AEs are symptoms or illnesses requiring a hospitalisation, or an emergency room visit, or visit to/by a health care provider.
Percentage of participants with SAEs, AEs leading to withdrawal, AESIs and medically attended AEs | During the 6 months (including the day of vaccination) following the second vaccination (Vaccine administered at Day 721)
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject or is an abnormal pregnancy outcome. AESIs are predefined (serious or non-serious) AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterise and understand it. Medically attended AEs are symptoms or illnesses requiring a hospitalisation, or an emergency room visit, or visit to/by a health care provider.

SECONDARY OUTCOMES:
Percentage of participants with hSBA titers ≥ LLOQ for N. meningitidis serogroups A, C, W and Y | At Baseline (Day 1), 1 month after the first dose of MenABCWY (Day 31) and 1 month after second dose of MenABCWY (Day 751 for the ABCWY-24 Group and Day 1471 for the ABCWY-48 Group)
  The immune response to 1 and 2 doses of the MenABCWY vaccine administered on a 0-, 24-month schedule, and a 0-, 48-month schedule is evaluated against N. meningitidis serogroups A, C, W and Y.
Percentage of participants with hSBA titers ≥ LLOQ for each N. meningitidis serogroup B indicator strains and for serogroups A, C, W and Y | At 25 months after the second dose of MenABCWY (Day 1471 for the ABCWY-24 Group)
  The antibody persistence at 25 months after the second dose of the MenABCWY vaccine administered on a 0-, 24-month schedule is evaluated against each N. meningitidis serogroup B indicator strains and serogroups A, C, W and Y.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (22):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Ventura, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Nicholasville, Kentucky
  - GSK Investigational Site, Haughton, Louisiana
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Layton, Utah
- Germany (6):
  - GSK Investigational Site, Bramsche
  - GSK Investigational Site, Herxheim
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Mannheim
  - GSK Investigational Site, Schönau am Königssee
  - GSK Investigational Site, Schweigen-Rechtenbach

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.